DOCUMENT

: Statistical Analysis Plan

DOCUMENT STATUS

: Final

PROJECT NO.

: 0110-23

STUDY IDENTIFIER

: 221030

An Open Label, Balanced, Randomized, Two-Treatment, Four-Period, Two-Sequence, Single Oral Dose, Full Replicate Crossover, Bioequivalence Study of Albendazole Tablets IP 400 mg of Biddle Sawyer Limited (GSK group company) with Albendazole Tablets 400 mg of Glaxo SmithKline Consumer Healthcare, South Africa (PTY) Ltd in Healthy, Adult Participants under Fed Condition.

SAP VERSION

: 00 (Based on Protocol version 1.0 dated 3<sup>rd</sup> July 2023)

SAP DATE

: 04 October 2023

SUPERSEDES

: None

**SPONSOR** 

: GSK Research & Development Limited,

980 Great West Road, Brentford, Middlesex, TW8 9GS, UK

PREPARED BY

: Lambda Therapeutic Research Limited,

Lambda house, Plot No. 38, Survey no. 388

Near Silver Oak Club, S. G. Highway,

Gota, Ahmedabad-382481,

Gujarat, India.

#### **CRO's SIGNATURES:**

| | Prepared<br>By | Prepared<br>by | Reviewed by | Approved by |
|---|---|---|---|---|
| Marsa | PPD | PPD | PPD | PPD |
| Name | M.Sc. | M.Sc. | M.Sc., M.Phil. | M.Sc. |
| Designation | Technical<br>Officer | Technical<br>Officer | Assistant General<br>Manager | PPD |
| Role | Biostatistician | SAS Programmer | Principal<br>Biostatistician | Head of the Department |
| Company's<br>Name | Lambda Therapeutic Research Ltd. | | | |
| Signature<br>& Date | PPD | | | |



## **SPONSOR'S SIGNATURE:**

| | Approved by |
|-------------------|-------------|
| Name | |
| Designation | |
| Organization Name | |
| Signature & Date | |



# INDEX

| AB | BREVIATIONS AND DEFINITIONS | 4 |
|-----|---------------------------------------------------------|------|
| 1 | Introduction | 6 |
| 2 | Objective, Endpoints and Estimands | 6 |
| 3 | Overall Study Design | 9 |
| 3.1 | Study Design | 9 |
| 3.2 | Study Intervention(s) Administered | 9 |
| | Sample Size | |
| 3.4 | Randomization | .11 |
| 3.5 | PK Sampling Schedule | .11 |
| 4 | Analysis sets | . 12 |
| 5 | Assessment of Pharmacokinetic Parameters | . 12 |
| 5.1 | Pharmacokinetic analysis | . 12 |
| | Pharmacokinetic Parameters | |
| 6 | Statistical Considerations | . 14 |
| 6.1 | Statistical Hypotheses | . 14 |
| | Multiplicity Adjustment | |
| | Statistical Analysis | |
| | 6.3.1 General considerations | |
| | 6.3.2 Primary Endpoint(s)/Estimand(s) Analysis | . 15 |
| | 6.3.2.1 Descriptive statistics | . 15 |
| | 6.3.2.2 Analysis of Variance (ANOVA) | |
| | 6.3.2.3 90% Confidence Interval | |
| | 6.3.2.4 Ratio analysis | |
| | 6.3.2.5 Intra-subject variability | |
| | 6.3.2.6 Missing and non-reportable values | |
| | 6.3.2.7 Intercurrent event and handling of missing data | |
| | 6.3.2.8 Bioequivalence criteria | |
| 7 | 6.3.3 Secondary Endpoint(s)/Estimand(s) Analysis | |
| 7 | Safety Assessment and Analysis | |
| | Safety Assessment | |
| | Safety Analysis | |
| | Change from the protocol | |
| | Interim analysis | |
| | Software Information for Analysis | |
| | Format Specifications for outputs | |
| | List of Tables | |
| | List of Listings | |
| | List of Figures | |
| | List of In-text Tables | |
| | Statistical Outputs | |
| | References | |
| 18 | Tables and Listings shells | .27 |

# ABBREVIATIONS AND DEFINITIONS

| λz | : | First order rate constant associated with the terminal (log-linear) |
|---|---|---|
| Abs | : | portion of the curve Absolute |
| ACE | : | Angiotensin converting enzyme |
| AE | : | Adverse event |
| ALT | : | Alanine aminotransferase |
| ANC | : | Absolute neutrophil count |
| ANOVA | : | Analysis of variance |
| AST | : | Aspartate aminotransferase |
| AUC | : | Area under the curve |
| AUC_%Extrap_obs | : | % Residual area |
| AUC0-∞ | : | Area under the plasma concentration versus time curve from time zero to infinity |
| AUC(0-t) | : | Area under the plasma concentration-time curve up to the last measured time point |
| BE | : | Bioequivalence |
| BMI | : | Body mass index |
| BSA | : | Body surface area |
| Cmax | : | Maximal (peak) plasma concentration |
| cm | : | Centimeter |
| CFB | : | Change from baseline |
| CI | : | Confidence interval |
| COVID | : | Corona virus disease |
| CV | : | Coefficient of variation |
| CRO | : | Contract research organization |
| ECG | : | Electrocardiogram |
| GMR | : | Geometric mean ratio |
| Hb | : | Hemoglobin |
| HBsAg | : | Hepatitis B surface antigen |
| HCV | : | Hepatitis C virus |
| НСТ | : | Hematocrit |
| HIV | : | Human immunodeficiency virus |
| h/hr/hrs | : | Hours |
| ICH | : | The international council for harmonisation of technical requirements for pharmaceuticals for human use |

| IP | : | Investigational product |
|---|---|---|
| kg | : | Kilograms |
| ln | : | Logarithmic value to the base 'e' |
| $m^2$ | : | Meter square |
| MCH | : | Mean cell hemoglobin |
| MCHC | : | Mean corpuscular hemoglobin concentration |
| MCV | : | Mean corpuscular volume |
| MedDRA | : | Medical dictionary for regulatory activities |
| mg | : | Milligram |
| min | : | Minimum |
| mL | : | Milliliter |
| NQ | : | Non-quantifiable |
| OTC | : | Over the counter medicine |
| PK | : | Pharmacokinetic(s) |
| PT | : | Preferred term |
| RBC | : | Red blood cell |
| RDW-CV | : | Red cell distribution width - coefficient of variation |
| R <sup>2</sup> | : | Goodness of fit statistic for the terminal phase, adjusted for the number of points used in the estimation of $\lambda z$ |
| SAE | : | Serious adverse event |
| SAP | : | Statistical analysis plan |
| SAS | : | Statistical analysis system |
| SD | : | Standard deviation |
| SGOT | : | Serum glutamic-oxaloacetic transaminase |
| SGPT | : | Serum glutamic pyruvic transaminase |
| SCABE | : | Scaled average bioequivalence |
| SOC | : | System organ class |
| SWR | : | Within-subject standard deviation of the reference study intervention |
| t1/2 | : | Terminal half-life |
| TOST | : | Two one-sided t-test |
| Tmax | : | Time of the maximum measured plasma concentration |
| WBC | : | White blood cell |
| WHO | : | World health organization |

#### 1 Introduction

This statistical analysis plan provides the framework for the analysis and summarization of the data generated from the study conducted to assess the bioequivalence Albendazole Tablets IP 400 mg (Test) of Biddle Sawyer Limited (GSK group company) compared with Albendazole Tablets 400 mg (Reference) of Glaxo SmithKline Consumer Healthcare, South Africa (PTY) Ltd in Healthy, Adult Participants under Fed Condition.

#### 2 Objective, Endpoints and Estimands

| Objectives | Endpoints |
|---|---|
| Primary | |
| To evaluate if Test Study Intervention (T): Albendazole tablets IP 400 mg, manufactured by Biddle Sawyer Limited is bioequivalent to Reference Study Intervention (R): Albendazole Tablets 400 mg, manufactured by GSK Consumer Healthcare, South Africa (PTY) | Albendazole Cmax and AUC(0-t) |
| Secondary | |
| To assess secondary pharmacokinetic parameters of Test Study Intervention (T): Albendazole tablets IP 400 mg relative to Reference Study Intervention (R): Albendazole tablets 400 mg. | <ul> <li>Albendazole AUC0-∞, Tmax, t1/2, lambda-z (λz) and AUC_%Extrap_obs.</li> <li>Albendazole sulfoxide Cmax, AUC(0-t), AUC0-∞, Tmax, t1/2, lambda-z (λz) and AUC_%Extrap_obs.</li> </ul> |
| To assess the safety and tolerability of<br>a single oral dose of the test versus the<br>reference study intervention. | <ul> <li>Incidence of AE.</li> <li>Absolute and change from baseline in vital signs parameters at each timepoint.</li> </ul> |

#### Primary estimand/coprimary estimands:

The primary clinical question of interest is:

To evaluate if Test Study Intervention (T): Albendazole tablets IP 400 mg is bioequivalent to Reference Study Intervention (R) Albendazole tablets 400 mg in healthy adult participants under fed conditions.

The estimand is described by the following attributes:



- **Population**: Healthy adult participants between 18 to 45 years of age.
- **Treatment condition**: Single dose of Albendazole tablets IP 400 or Albendazole tablets 400 mg, each treatment period given under fed conditions to healthy participants.
- Variable/endpoint: Cmax and AUC(0-t)

#### • Summary measure:

o Treatment ratios of geometric least square means with 90% CI, and within-subject coefficient of variation of reference study intervention (intra-subject CV in %).

#### • Intercurrent events:

- Permanent Treatment discontinuation due to any reason (includes COVID-19 positive, AE related withdrawal etc.) While-on treatment strategy that is, all available data up until the withdrawal of the consent will be reported.
- Use of prohibited or rescue medication which could affect PK parameters (Cmax and AUC(0-t)) during the study - Hypothetical strategy
- Experiences emesis/vomiting before 2 times of median Tmax (i.e. 2 x 2hour = 4hour) after dose administration - Hypothetical strategy.

#### • Rationale for estimand:

- o The rationale of the while on treatment strategy is to estimate the PK parameters when participants have taken the dose/treatment condition.
- The rationale of hypothetical strategy for prohibited/rescue medication is to minimize the potential confounding of PK data (Cmax and AUC(0-t)). It attempts to estimate treatment effects had the intercurrent event not occurred. In this scenario, if the intercurrent event occurred before 2 times median Tmax (i.e. 2 x 2hour = 4hour) after study drug administration, PK parameters (Cmax and AUC (0-t)) data would be set to be missing for that period.
- o Hypothetical strategy would be considered if emesis/vomits occur before 2 times the median Tmax (i.e., 2 x 2hour = 4hour) after study drug administration in particular period, this is because the drug would not have been absorbed into the body. In this situation, PK parameters (Cmax and AUC(0-t)) data would set to be missing for that period.

#### Secondary estimand(s) - PK endpoint

The secondary clinical question of interest is:

To assess secondary pharmacokinetic parameters of Test Study Investigation (T): Albendazole tablets IP 400 mg relative to Reference Study Investigation (R): Albendazole tablets 400 mg.

The estimand is described by the following attributes:

- **Population**: Healthy adult participants between 18 to 45 years of age.
- •Treatment condition: Single dose of Albendazole tablets IP 400 mg or Albendazole tablets 400 mg, each treatment period given under fed conditions to healthy participants.

#### Variable/endpoint:

- Albendazole AUC0- $\infty$ , Tmax, t1/2,  $\lambda z$  and AUC %Extrap obs.
- Albendazole sulfoxide Cmax, AUC(0-t), AUC0-∞, Tmax, t1/2, λz and AUC %Extrap obs.

#### **Summary measure:**

Descriptive statistics (N, n, arithmetic mean, 95% CI of arithmetic mean, SD, median, minimum, maximum, and geometric mean) will be presented for untransformed secondary PK parameters (AUC0- $\infty$ , AUC(0-t), Tmax, t1/2,  $\lambda$ z and AUC\_%Extrap\_obs).

#### • Intercurrent events:

Same as primary endpoint

#### Rationale for estimand:

o The rationale of hypothetical strategy which is impacted to secondary PK parameters (AUC0-∞, AUC(0-t), Tmax, t1/2, λz and AUC\_%Extrap\_obs) during the study is same as primary estimands.

#### **Secondary estimand(s) - 2(Safety)**

The secondary clinical question of interest is:

To assess the safety and tolerability of a single oral dose of Test Study Intervention (T): Albendazole tablets IP 400 mg relative to Reference Study Intervention (R): Albendazole tablets 400 mg.

The estimand is described by the following attributes:

- **Population**: Healthy adult participants between 18 to 45 years of age.
- **Treatment condition**: Single dose of Albendazole tablets IP 400 mg or Albendazole tablets 400 mg, each treatment period given under fed conditions for healthy participants.
- Variable/endpoint: Incidence of AE and Absolute and change from baseline in vital signs parameters at each timepoint.

#### • Summary measure:

- o Number and percentage will be presented for incidence of AE.
- o Descriptive statistics (N, n, mean, SD, median, minimum, and maximum) will be presented for absolute and change from baseline values of vital signs parameters at each timepoint.

#### • Intercurrent events:

Permanent Treatment discontinuation due to any reason (includes COVID-19 positive, AE related withdrawal etc.) - Treatment policy strategy.

#### • Rationale for estimand:

Permanent Treatment discontinuation due to any reason will be handled with a treatment policy strategy as occurrence of AE until participant are on study will be collected and reported.

#### 3 Overall Study Design

#### 3.1 Study Design

An Open Label, Balanced, Randomized, Two-Treatment, Four-Period, Two-Sequence, Single Oral Dose, Full Replicate Crossover, Bioequivalence Study of Albendazole Tablets IP 400 mg of Biddle Sawyer Limited (GSK group company) with Albendazole Tablets 400 mg of GSK Consumer Healthcare, South Africa (PTY) Ltd in Healthy, Adult Participants under Fed Condition.

Based on , this study will employ 2 sequences in a 4-period cross-over design, i.e. T-R-T-R and R-T-R-T (T=test study intervention, R=reference study intervention).

#### Study design overview



#### 3.2 Study Intervention(s) Administered

| Intervention Label | Test (T) | Reference (R) |
|---|---|---|
| Intervention Name | Albendazole tablets IP 400 mg | Albendazole 400 mg tablets |
| <b>Intervention Description</b> | Solid dosage form | Solid dosage form |
| Type | Drug | Drug |
| Dose Formulation | Tablet | Tablet |
| Unit Dose Strength(s) | 400 mg | 400 mg |
| Dosage Level(s) | single oral dose of 400 mg | single oral dose of 400 mg |
| Route of Administration | oral | oral |
| Use | active comparator | active comparator |
| IMP and NIMP/AxMP. | Study intervention | Study intervention |
| Sourcing | Provided by the sponsor | Provided by the sponsor |
| Packaging and Labeling | Study intervention will be provided in container. Each container will be labeled as required per country requirement. | Study intervention will be provided in container. Each container will be labeled as required per country requirement. |

#### 3.3 Sample Size

Based on the WHO guideline for albendazole, the maximum intra-subject variability observed for primary pharmacokinetic parameters Cmax and AUC(0-t) could be up to  $\sim 68\%$  and 62% respectively. For this sample size calculation, a product difference of up to 10% (i.e. T/R ratio as 90.0-111.1%) has been assumed.

The sample size was determined using R software considering the following assumptions:

- a. T/R ratio = 90.0-111.1%
- b. Intra-Subject CV (%)  $\sim 68\%$  (Cmax) and 62% (AUC(0-t)), or 48% (both)
- c. Significance Level = 5%

Correlation between Cmax and AUC(0-t) was calculated to be very high, based on an in-house albendazole study (GSK study O7921353). The exact Cmax and AUC(0-t) covariance matrix was calculated from this historical study as per below table and used to simulate realistic Cmax and AUC(0-t) values based on multivariate normal distributions. These values were then used to perform joint power calculation on the basis of inclusion of 70 participants with varying levels of missing data. To determine the power, success rates were based on 1000 replicates of the study design.

Table 1 Covariance matrix used for Cmax and AUC(0-t) in power calculations

| | AUC(0-t) | Cmax |
|--------------------|----------|-------|
| AUC <sub>0-t</sub> | 0.814 | 0.685 |
| Cmax | 0.685 | 0.747 |

Table 2 Joint power calculation results (N=1000) across various scenarios of missing data

| Scenario | Joint Power (CV% = 48% for both Cmax and | Joint Power (CV% = 68% and 62% for AUC(0-t) and |
|---|---|---|
| | AUC(0-t) | Cmax respectively) |
| 48 participants have complete data for Cmax and AUC(0-t) for all 4 periods and 22 Participants data is completely missing | 90.3% | 93.7% |
| 48 participants have complete data for Cmax and AUC(0-t) for all 4 periods, 10 participants have 2 period data and 12 participants data is completely missing | 93.4% | 95.8% |
| 48 participants have complete data for Cmax and AUC(0-t) for all 4 periods, 6 participants have data for 2 periods and 16 remaining participants have no data at all | 91.5% | 94.9% |

Based on these results, and the aforementioned covariance matrix, at least 48 participants would be required to power a study to 90% to establish bioequivalence under the assumptions



highlighted above. Based on experience, ~30% dropouts and/or withdrawals (due to unavoidable reasons like medical ground, adverse events, own accord, etc.) should be considered, requiring a target inclusion of 70 participants for this study. In-house data showed the variance of Cmax and AUC to be closer to 48%, implying that the above sample size calculation takes into account the worst-case scenario, and may in fact provide a power of > 95%.

Sufficient number of volunteers will be asked to report on the day of check-in of period I in order to ensure that at least **70 participants** will be enrolled in the beginning of the study. Subsequent dropouts after dosing in period I will not be replaced.

**Note:** Additional participants if available, may be checked-in on the day of check in of period I to compensate for any dropout prior to dosing of period I. These participants will be dosed if there are dropouts prior to dosing in period I. If there are no dropouts, these participants will be checked-out without being dosed after completion of dosing in period I.

#### 3.4 Randomization

Participants will be assigned either of the two sequence 'TRTR' or 'RTRT' based on the randomization schedule by Lambda generated using SAS® Version 9.4 or higher (SAS Institute Inc., USA). Equal allocation of participants in each sequence is planned.

The personnel involved in dispensing of study intervention and verification of dispensed study interventions will be accountable for ensuring compliance to randomization schedule.

#### 3.5 PK Sampling Schedule

A total of 22 blood samples each of 3 mL, will be collected from each participant in each period.

The venous blood samples will be withdrawn at the following times. All actual sample times will be recorded in addition to their planned time.

| | Time neints | Proposed clock time | Analytes to | Analytes to measure |
|---|---|---|---|---|
| Day | Time points<br>(Hours) | | Albendazole | Albendazole<br>Sulfoxide |
| | Pre-dose (0.00) | Within 60 minutes prior to dosing | √ | V |
| | 0.33 | 0h20min | <b>√</b> | V |
| _ | 0.67 | 0h40min | $\sqrt{}$ | V |
| | 1.00 | 1h00min | √ | V |
| _ | 1.33 | 1h20min | √ | V |
| 1 | 1.67 | 1h40min | $\sqrt{}$ | V |
| | 2.00 | 2h00min | $\sqrt{}$ | V |
| | 2.33 | 2h20min | $\sqrt{}$ | V |
| _ | 2.67 | 2h40min | √ | V |
| | 3.00 | 3h00min | √ | V |
| | 3.33 | 3h20min | √ | V |
| | 3.67 | 3h40min | V | V |
| | 4.00 | 4h00min | V | V |

| | Time points<br>(Hours) | Proposed clock time | Analytes to measure | |
|---|---|---|---|---|
| Day | | | Albendazole | Albendazole<br>Sulfoxide |
| | 4.50 | 4h30min | √ | V |
| | 5.00 | 5h00min | V | V |
| | 6.00 | 6h00min | V | V |
| | 8.00 | 8h00min | V | V |
| | 10.00 | 10h00min | √ | V |
| | 12.00 | 12h00min | √ | $\sqrt{}$ |
| | 14.00 | 14h00min | √ | V |
| 2 | 18.00 | 18h00min | V | V |
| | 24.00 | 24h00min | √ | V |

Day 1: Day of study intervention administration in each period.

#### 4 Analysis sets

The analysis set will be defined as follows:

| Analysis<br>Sets | Description | Analysis Evaluate |
|---|---|---|
| Randomized | All participants assigned to study treatment | Study Population |
| Safety set | The safety set will include all randomized participants who receive at least 1 dose of study medication. The safety population will be used for all analyses of safety data. | Safety |
| PK set | All participants in the Safety set who had at least 1 measurable PK assessment (for the purpose of the PK analysis, only those participants in this dataset who have evaluable data for one test and one reference period will be used). | PK |

#### 5 Assessment of Pharmacokinetic Parameters

#### 5.1 Pharmacokinetic analysis

Pharmacokinetic analysis will be performed on the available concentration data of all the participants.

Criteria for exclusion of pharmacokinetic parameters of particular participants from statistical analysis will be as below:

Participants who were discontinued/withdrawn and do not have evaluable data for at least 1 treatment and 1 reference drug period will be excluded.

Day 2: Subsequent day after study intervention administration in each period.

Three consecutive missing (M) / Non-Reportable (NR) samples in elimination phase may significantly influence the AUC(0-t) and elimination phase dependent parameters (AUC0- $\infty$ , AUC0-t, t1/2,  $\lambda z$ , AUC\_%Extrap\_obs). Inclusion of such parameters in the statistical analysis may mislead the final outcome. Hence, AUC(0-t) and elimination phase dependent parameters (AUC0- $\infty$ , AUC(0-t), t1/2,  $\lambda z$ , AUC %Extrap obs) will be excluded.

The concentration—time profiles of subjects who exhibit pre-dose concentrations higher than 5% of the corresponding Cmax of that period will be excluded from the statistical analysis [Note: a statistical sensitivity analysis including the same will be provided for information purpose].

Participants without measurable concentrations or who have only very low plasma concentrations relative to that of the product in question, will be excluded from the pharmacokinetic and statistical analyses. A participant is considered to have very low plasma concentrations if their AUC is less than 5% of the geometric mean AUC of the product in question, calculated without inclusion of data from the outlying participant [Note: statistical analysis with including the same will be provided for information purpose].

Note: This exclusion will be period specific.

#### **5.2 Pharmacokinetic Parameters**

The following pharmacokinetic parameters will be computed for albendazole and albendazole sulfoxide using non-compartmental model of Phoenix<sup>®</sup> WinNonlin<sup>®</sup> Version 8.3 or higher (Certara L.P.) for each period:

• Primary Pharmacokinetic Parameters: Cmax, AUC<sub>0-t</sub>

• Secondary Pharmacokinetic Parameters: AUC<sub>0-∞</sub>, Tmax, λz, t1/2, AUC %Extrap obs

| Primary PK Paran | net | ers: |
|---|---|---|
| Cmax | : | Maximum measured plasma concentration. |
| AUC(0-t) | •• | Area under the plasma concentration versus time curve from time zero to the last measurable concentration as calculated by linear trapezoidal method. |
| Secondary PK Par | am | neters |
| AUC0-∞ | : | Area under the plasma concentration versus time curve from time zero to time infinity. Where $AUC0-\infty = AUC(0-t) + Ct/\lambda z$ , Ct is the last measurable concentration and $\lambda z$ is the terminal rate constant. |
| Tmax | : | Time of the maximum measured plasma concentration. |
| λz | : | First order rate constant associated with the terminal (log-linear) portion of the curve. This is estimated via linear regression of time vs. log concentration. This parameter will be calculated by linear least squares regression analysis using at least last 3 non-zero plasma concentration values. |
| t1/2 | : | The terminal half-life will be calculated as 0.693/λz. |
| AUC_%Extrap_obs | : | The residual area in percentage will be determined by the formula, $[(AUC0-\infty - AUC0-t)/AUC0-\infty] \times 100$ . |

For all the above computations, actual time points of the sample collection will be used.

Non-quantifiable (NQ) data, such as concentrations below the quantification limit may be excluded or omitted, depending on where they are located in time, see Section 6.3.2.6.

No value of  $\lambda_z$ , AUC<sub>0-∞</sub>, AUC\_%Extrap\_obs and  $t_{1/2}$  will be reported for cases that do not exhibit a terminal log-linear phase in the concentration versus time profile.

#### 6 Statistical Considerations

#### 6.1 Statistical Hypotheses

According to WHO product specific guidance (Notes on the Design of Bioequivalence Study: Albendazole; 29 March 2021), albendazole pharmacokinetics in the fed state is highly variable (up to 68% for Cmax and 62% for AUC). Therefore, this study was designed as a replicate cross-over study, to estimate variability more accurately and, if indicated, to widen the acceptance range for Cmax and AUC(0-t) (, 2021). Considering the same, full replicate study has been planned in line with WHO product specific guidance document and reference-scaled average bioequivalence approach will be used for hypothesis testing.

The null hypothesis to be tested is:

$$H_0: \frac{\left(\mu_T - \mu_R\right)^2}{\sigma_{WR}^2} \ge \ \theta$$

Versus alternative hypothesis

$$H_1: \frac{\left(\mu_T - \mu_R\right)^2}{\sigma_{WR}^2} < \theta$$

Where:  $\mu_T$  and  $\mu_R$  are the means of ln-transformed PK parameters (Cmax and/or AUC) obtained from the BE study for the test and reference products, respectively.

 $\sigma_{WR}$  is the within-subject standard deviation of the ln-transformed values of PK parameter of the reference study intervention.

Testing will be performed at a level of 0.05 and  $\theta$  is the scaled average BE limit.

The test drug must pass for primary endpoint PK parameters (Cmax and AUC(0-t)) to demonstrate BE to the reference drug. Let  $\sigma_{W0}$  be the regulatory constant (based on 0.80-1.25 geometric mean ratio restriction criteria) and assumed to be 0.294.

a. The 90% confidence interval of GMR of T/R must be contained within [U, L] = exp [ $\pm k \cdot s_{WR}$ ], which is scale acceptance limit based on k( $\theta S$ ),

Where  $k = \ln(1.25)/\sigma_{W0}$  which is approx. 0.760

U is the upper limit of the acceptance range, L is the lower limit of the acceptance range,  $s_{WR}$  is the within-subject standard deviation of the ln-transformed values of PK parameter of the reference study intervention.

b. Point estimate of GMR of T/R should be between 80.00 –125.00%.

For the parameters Cmax and AUC(0-t), if the intra-subject  $CV_W$  of for the reference study intervention is less than or equal to 0.30 upon trial completion for any of these treatment group, conventional average BE approach with TOST procedure with  $\alpha$ =0.05 for each one-sided test will

## Albendazole Tablets IP 400 mg

be used to test  $0.8 \le GMR \le 1.25$ . This is equivalent to requiring that a 90% interval for the true ratio of test to reference geometric means falls entirely within the range of 80.00 to 125.00%. If the intra-subject coefficient of variation (CV<sub>W</sub>) of for the reference study intervention is greater than 0.30 upon trial completion, a reference-scaled average bioequivalence approach will be used<sup>3</sup>.

If the intra-subject variability for Cmax and AUC(0-t) following replicate administrations of the comparator product is > 30%, the acceptance criteria for Cmax and AUC(0-t) will be widened to a maximum of 69.84–143.19%.

#### 6.2 Multiplicity Adjustment

No multiplicity adjustment is required for this bioequivalence study.

#### 6.3 Statistical Analysis

#### **6.3.1** General considerations

The pharmacokinetic parameters will be analyzed to evaluate the differences between the test and reference study interventions by applying referenced scaled average bioequivalence approach. This approach will be assessed based on GMR and 90% confidence interval for ln-transformed PK parameters Cmax and AUCt using RSABE.

All the statistical analysis will be performed using SAS® Version 9.4 or higher (SAS Institute Inc., USA).

The participants having pharmacokinetic parameters available for 2 reference treatments will be included for calculation of intra-subject variability of reference study intervention.

Descriptive statistics & average bioequivalence analysis will be performed on the participants having pharmacokinetic parameters available for at least 1 test and 1 reference arm.

#### 6.3.2 Primary Endpoint(s)/Estimand(s) Analysis

#### **6.3.2.1** Descriptive statistics

Statistical analysis for primary endpoints will include descriptive statistics for the following pharmacokinetic parameters:

Cmax and AUC(0-t)

Descriptive statistics (N, n, arithmetic mean, 95% CI of arithmetic mean, geometric mean, 95% CI of geometric mean, SD, median, minimum and maximum) will be presented for primary PK parameters.

Average values of Test Study Intervention-T and Reference Study Intervention-R for PK parameters for each participant will be calculated and reported. Descriptive statistics will be calculated and reported for the same data.

Individual values of PK parameters for Test Study Intervention-T (first administration), Test Study Intervention-T (second administration), Reference Study Intervention-R (first administration) and Reference Study Intervention-R (second administration) for each participant will be calculated and reported. Descriptive statistics will be calculated and reported for the same data.

Version 00



PK parameters will be analyzed to evaluate the differences between the test and reference products by applying SCABE following EMA guidelines in investigation of bioequivalence regarding highly variable drug product (% of CVw >30), otherwise ABE will be applied.

#### 6.3.2.2 Analysis of Variance (ANOVA)

Analysis of Variance (ANOVA) will be used on ln-transformed pharmacokinetic parameters Cmax and AUC(0-t) for albendazole or albendazole sulfoxide. The ANOVA model will include sequence, participant(sequence), period and formulation as fixed effects.

Each analysis of variance will include calculation of ratio of geometric least-squares means and the standard error associated with these ratios.

The above statistical analyses will be done using PROC GLM of SAS® procedure. A significance level of 5% (alpha =0.05) will be used for the model.

#### 6.3.2.3 90% Confidence Interval

90% confidence intervals for the ratio of geometric least squares means between drug formulations will be calculated for ln-transformed data of Cmax and AUC(0-t) for albendazole and albendazole sulfoxide.

#### 6.3.2.4 Ratio analysis

Ratio of geometric least squares means of test and reference formulations will be computed and reported for ln-transformed pharmacokinetic parameters Cmax and AUC(0-t) for albendazole and albendazole sulfoxide.

#### 6.3.2.5 Intra-subject variability

Intra-subject variability of reference study intervention-R will be computed and reported for Intransformed pharmacokinetic parameters Cmax and AUC(0-t) for albendazole and albendazole sulfoxide.

The existence of outlier subjects that inflate the intra-subject variability will be assessed. In case of such outliers, results will be reported with and without those outliers.

#### 6.3.2.6 Missing and non-reportable values

If 1 or more NQ values occur in a profile before the first measurable concentration, they will be assigned a value of zero concentration.

If a single NQ value occurs between measurable concentrations in a profile, the NQ should be omitted (set to missing) in the derivation of pharmacokinetic parameters and statistical analysis.

If 2 or more NQ values occur in succession between measurable concentrations, the values in question will be set to missing. For the derivation of pharmacokinetic parameters, these NQs will be omitted. The NQ values will be set to 0 and the trapezoidal rule will be applied to all the observed data.

NQs which occur after the last measurable concentration will be omitted (set to missing) in the derivation of pharmacokinetic parameters and statistical analysis. Any missing samples (M) concentration value will be disregarded in pharmacokinetic and statistical analysis.

#### 6.3.2.7 Intercurrent event and handling of missing data

The data will be affected by occurrence of the intercurrent event and only data available while the participant is receiving the treatment will be used under while-on treatment policy strategy. Participant level missing data will not be imputed, and available data will be used in the analysis.



In the case of emesis/vomiting or use of prohibited/rescue medication, the data for that period will not be used for the analysis of PK parameters relating to the primary endpoint using hypothetical strategy.

#### 6.3.2.8 Bioequivalence criteria

Based on the statistical results of 90% confidence interval for the ratio of the geometric least square means for both ln-transformed pharmacokinetic parameters Cmax and AUC(0-t), conclusion will be drawn for Test Study Intervention-T vs. Reference Study Intervention-R for albendazole with following considerations.

#### For Cmax and AUC(0-t):

- 1. If within-reference intra-subject CV of ln-transformed Cmax and/or AUC(0-t)  $\leq$  30% then bioequivalence of the test study intervention with that of the reference study intervention will be concluded, if the 90% confidence interval falls within the acceptance range of 80.00–125.00% for ln-transformed pharmacokinetic parameter Cmax and AUC(0-t).
- 2. If within-reference intra-subject CV of ln-transformed Cmax and/or AUC(0-t) > 30% then Cmax and/or AUC(0-t) limit will be widened using scaled-average-bioequivalence. Under scaled-average-bioequivalence, [U,L] = exp [ $\pm k \cdot _{SWR}$ ] where U is the upper limit of the acceptance range, L is the lower limit of the acceptance range, k is the regulatory constant set to 0.760 and  $S_{WR}$  is the within-subject standard deviation of the ln transformed values of Cmax and/or AUC(0-t) of the reference study intervention.
- 3. If within-reference intra-subject CV of ln-transformed Cmax and/or AUC(0-t)  $\geq$  50% then Cmax and/or AUC(0-t) bioequivalence limits will be widened to a maximum of 69.84 143.19%.

Bioequivalence of the test study intervention with that of the reference study intervention will be concluded for Cmax and AUC(0-t), if both of the following conditions are satisfied:

- The 90% confidence interval for ln-transformed data of Cmax and AUC(0-t) falls within the respective newly widen range [U, L] =  $\exp\left[\pm k \cdot _{SWR}\right]$ , which is based upon the within-subject variability observed for respective pharmacokinetic parameter.
- The geometric least square mean ratio (GMR) of test to reference for Cmax and AUC(0-t) falls within the acceptance range of 80.00–125.00%.

Data of metabolite albendazole sulfoxide will be provided as supportive information only.

#### 6.3.3 Secondary Endpoint(s)/Estimand(s) Analysis

Statistical analysis for secondary endpoints will include descriptive statistics for the following pharmacokinetic parameters:

Albendazole: AUC0-∞, Tmax, t1/2, λz and AUC %Extrap obs

Albendazole sulfoxide: AUC0-∞, AUC0-t, Cmax, Tmax, t1/2, λz and AUC %Extrap obs.

Descriptive statistics (N, n, arithmetic mean, 95% CI of arithmetic mean, SD, median, minimum, maximum and geometric mean with 95% CI) will be presented for untransformed secondary PK parameters.

Average values of Test Study Intervention-T and Reference Study Intervention-R for PK parameters for each participant will be calculated and reported. Descriptive statistics will be calculated and reported for the same data.

Individual values of PK parameters for Test Study Intervention-T (first administration), Test Study Intervention-T (second administration), Reference Study Intervention-R (first administration) and Reference Study Intervention-R (second administration) for each participant will be calculated and reported. Descriptive statistics will be calculated and reported for the same data.

In case of treatment discontinuation due to any reason, only the data available before the occurrence of intercurrent event will be used to estimate secondary PK parameters using while-on-treatment policy strategy.

If any participant experience emesis/vomiting or if a prohibited/rescue medication is used by any participant, the participant's data for that period will not be used for the analysis of secondary endpoints related to PK using hypothetical strategy.

Treatment policy strategy will be used to analyze the secondary endpoints related to safety to make use of all available data for a participant.

#### 7 Safety Assessment and Analysis

#### 7.1 Safety Assessment

#### Demographic data

Demographic data such as date of birth, sex, race, age, and ethnicity will be assessed on screening visit.

#### **Body Measurement**

Body measurement data such as height, weight and BMI will be assessed on screening visit.

#### **Medication history**

Current medication (prescribed medication & OTC medication, herbal remedies, cimetidine, praziquantel, dexamethasone, ritonavir, phenytoin, carbamazepine, phenobarbital) and usage of any concomitant therapy or any ingestion of medicine in the previous 14 days prior to dosing of period I and any vaccine (including COVID-19 vaccine) from 14 days prior to dosing of period I. Medication history will be recorded on PERIOD 1 (Day 1)

#### Physical examination

Physical examination will be assessed on screening visit, check in (Day 1) and check-out (Day 2) of each period.

#### Urine drug scan and breath alcohol test

Drug abuse in urine and Breath alcohol test will be performed on check-in of each period.

#### Chest X-ray

Chest X-ray (within the last 6 months) (postero-anterior view) will be carried out at the time of screening.

#### Vital signs

Vitals (sitting blood pressure and radial pulse) will be recorded at pre-dose (within 60 minutes before the dosing) and at 2, 4, 6, 12 and 24 hours post-dose in each period.

Note: All post-dose vitals will be performed within  $\pm$  40 minutes of the scheduled time.

Recording of vital signs (blood pressure, respiratory rate and radial pulse and body temperature) will be done at screening, after check-in, before check-out in each period.



Note: Vital signs before checkout may be started 120 minutes prior to the scheduled time of checkout of each participant.

#### 12-lead ECG

12-lead ECG will be carried out at the time of screening (up to 28 days before Dosing in period I).

#### Clinical safety laboratory tests

Serology tests (HIV AB (1 & 2), Anti HCV and HBsAg) will be performed at the time of screening. Urine parameters will be performed at the time of screening.

<u>Urine parameters</u>: Specific Gravity, Leucocytes, Bilirubin, Urobilinogen, Erythrocytes, pH, Protein, Ketones, Glucose, Nitrite, Microscopic examination (As applicable).

Laboratory assessment for hematology and biochemistry will be performed at the time of screening. Laboratory assessment for hematology and biochemistry (except random glucose, sodium, potassium, chloride, alkaline phosphatase) will be performed at the end of the study (at the time of check-out of period IV).

Laboratory assessment for liver function test (SGPT, SGOP and total bilirubin) will be performed prior to check-in of period II, III and IV.

<u>Hematology</u>: Hemoglobin [Hb], RBC count, HCT, MCV, MCH, MCHC, RDW CV, Platelet count, WBC (total), Neutrophils %, Lymphocytes %, Eosinophils %, Monocytes %, Basophils %, Neutrophils abs, Eosinophils abs

<u>Biochemistry</u>: Random Glucose, Bilirubin Total, Total Protein, Albumin, Serum Globulin, A/G ratio, SGOT (AST), SGPT (ALT), Creatinine, Blood Urea Nitrogen, Sodium, Potassium, Chloride, Alkaline phosphatase.

#### **Pregnancy testing**

Serum Pregnancy test for female participants will be done at the time of screening, prior to checkin of each period and at the end of the study (at the time of check-out of period IV). Pregnancy testing must be done even if the participant is menstruating at the time of the study visit. The study intervention may only be administered if the pregnancy test is negative.

#### 7.2 Safety Analysis

Safety analysis will be done on the safety set. Safety variables include AEs, clinical laboratory parameters, vital signs, physical examinations. Safety variables will be listed and summarized with descriptive statistics as appropriate.

Continuous variables will be Summarized by treatment/sequence group using summary statistics (number of observations, mean, standard deviation, median, minimum and maximum etc.) as applicable. Categorical values will be summarized by the treatment group using frequencies and percentages.

Result obtained when evaluating safety (adverse events, vital signs, clinical laboratory tests etc.) will be listed and evaluated descriptively.

#### Adverse events

All AEs reported during the study must be included in the safety analysis. AEs will be classified by system organ class, by preferred term from the MedDRA version 25.0 or higher. They will be presented in individual listings and summary tables, and evaluated descriptively and in terms of



frequencies, by treatment. As will be summarized for all subjects in Safety set across two treatment groups by System Organ Class (SOC) and Preferred Term (PT). p-value using chi-square test or fisher exact test will be provided for the AE data.

Intensity refers to the severity of the AE.: Mild, Moderate, Severe.

#### Clinical laboratory values

LAMBDA

Clinical laboratory values will be compared to their reference ranges. Values outside the normal ranges will be highlighted. The Investigator has to comment, whether the abnormality is clinically relevant.

#### Other safety parameters

All results of vital sign measurements will be presented in individual listings. Where appropriate, results and possible changes in parameters will be evaluated descriptively or by descriptive statistics (mean, SD, median, range). Descriptive statistics (N, n, mean, SD, median, minimum and maximum) will be presented for absolute and change from baseline values of vital signs parameters at each timepoint.

Demographic data will be shown in tables as mean values, SD and ranges (min, max).

Clinical laboratory data will be shown in tables as mean values, SD and ranges (min, max) as applicable.

Physical examination, 12 lead ECG, Chest X-Ray performance and concomitant medication will be presented in data listings.

#### **Protocol deviations**

A list of all protocol deviations and an assessment of their impact will be included in listing. The deviations will include dosing related, IMP related, lab related, early, late or missed safety assessments, etc.

A number of participants with minor and major deviations will be provided.

#### 8 Change from the protocol

"The ANOVA model will include sequence, participant(sequence), period and formulation as fixed effects" as per the WHO requirements.

#### 9 Interim analysis

No interim analysis has been planned in this study.

#### 10 Software Information for Analysis

SAS® Version 9.4 or higher (SAS Institute Inc., USA) will be used for statistical and safety analysis.

Phoenix® WinNonlin® Version 8.3 or higher (Certara L.P.) will be used for pharmacokinetic analysis.

#### 11 Format Specifications for outputs

1. Output files of SAS procedures/Phoenix WinNonlin (statistical analyses, summary tables, individual data listings, etc.) will be produced as PDF files.



Project No. 0110-23 Version 00

- 2. Each individual PDF file will contain the statistical analysis output, i.e. a summary table, or data listing grouped by treatment or/and visit, for one analysis population, and for a single type of analysis.
- 3. The rules for grouping may vary according to the type of data (study outcome, safety), individual data listings, listings of derived variables, etc. and the type of output file which is produced (statistical analyses, summary tables, graphs).
- 4. Page format will be "A4".
- 5. Each listing will be numbered in the format Page X of Y (where Y denotes total number of pages in that particular listing). Page number will appear in the bottom right part of the listing.
- 6. For each output, 'Lambda Therapeutic Research Ltd.' Will appear in the Top left corner of the Header, 'Confidential' and 'Title' of the output will appear in the Centre of the Header and towards the Top right corner the 'project number' will be presented.
- 7. The font and font size for header/footer and body of the output will be Courier New size 9 pt which will be generated from SAS. The font and font size for header/footer and body of the output will be Times New Roman 12 pt which will be generated from Phoenix WinNonlin.

# 12 List of Tables

| 14.1 | Demographic data |
|---|---|
| 14.1.1 | Demographic data and baseline characteristics (Randomized set) |
| 14.1.2 | Demographic data and baseline characteristics (Safety set) |
| 14.1.3 | Demographic data and baseline characteristics (PK set) |
| 14.1.4 | Visit wise distribution of subjects (Randomized set) |
| 14.1.5 | Visit wise distribution of subjects (Safety set) |
| 14.1.6 | Visit wise distribution of subjects (PK set) |
| 14.1.7 | Summary of protocol deviations |
| 14.2 | Pharmacokinetic data |
| 14.2.1 | Plasma albendazole data |
| 14.2.1.1 | Summary statistics of pharmacokinetic parameters for albendazole |
| 14.2.1.2 | Pharmacokinetic parameters (untransformed) of albendazole for Test Product-T and Reference Product-R |
| 14.2.1.3 | Individual pharmacokinetic parameters (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration) |
| 14.2.1.4 | Pharmacokinetic parameters (untransformed) of data excluded from statistical analysis for albendazole (if applicable) |
| 14.2.1.5 | Pharmacokinetic parameters (ln-transformed) of albendazole for Test Product-T and Reference Product-R |
| 14.2.1.6 | Individual pharmacokinetic parameters (In-transformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration) |
| 14.2.1.7 | Plasma concentration of albendazole for Test Product-T1 (first administration) |
| 14.2.1.8 | Plasma concentration of albendazole for Test Product-T2 (second administration) |
| 14.2.1.9 | Plasma concentration of albendazole for Reference Product-R1 (first administration) |
| 14.2.1.10 | Plasma concentration of albendazole for Reference Product-R2 (second administration) |
| 14.2.1.11 | Plasma concentration of data excluded from statistical analysis for albendazole (if applicable) |
| 14.2.2 | Plasma albendazole sulfoxide data |
| 14.2.2.1<br>14.2.2.2 | Summary statistics of pharmacokinetic parameters for albendazole sulfoxide<br>Pharmacokinetic parameters (untransformed) of albendazole sulfoxide for Test |
| 14.2.2.3 | Product-T and Reference Product-R<br>Individual pharmacokinetic parameters (untransformed) of albendazole<br>sulfoxide for Test Product-T1 (first administration), Test Product-T2 (second<br>administration), Reference Product-R1 (first administration) and Reference<br>Product-R2 (second administration) |





| 14.2.2.4 | Pharmacokinetic parameters (untransformed) of data excluded from statistical analysis for albendazole sulfoxide (if applicable) |
|---|---|
| 14.2.2.5 | Pharmacokinetic parameters (In-transformed) of albendazole sulfoxide for Test<br>Product-T and Reference Product-R |
| 14.2.2.6 | Individual pharmacokinetic parameters (ln-transformed) of albendazole sulfoxide for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration) |
| 14.2.2.7 | Plasma concentration of albendazole sulfoxide for Test Product-T1 (first administration) |
| 14.2.2.8 | Plasma concentration of albendazole sulfoxide for Test Product-T2 (second administration) |
| 14.2.2.9 | Plasma concentration of albendazole sulfoxide for Reference Product-R1 (first administration) |
| 14.2.2.10 | Plasma concentration of albendazole sulfoxide for Reference Product-R2 (second administration) |
| 14.2.2.11 | Plasma concentration of data excluded from statistical analysis for albendazole sulfoxide (if applicable) |
| 14.2.3 | Actual time points used for pharmacokinetic evaluation |
| 14.3 | Safety data |
| 14.3.1 | Overall summary of treatment emergent adverse events (Safety set) |
| 14.3.2 | Summary of treatment emergent adverse events by system organ class and preferred term (Safety set) |
| 14.3.3 | Summary of treatment emergent adverse events by relationship to study drug and system organ class and preferred term (Safety set) |
| 14.3.4 | Summary of treatment emergent adverse events by severity grade and system organ class and preferred term (Safety set) |
| 14.3.5 | Summary of subject disposition |
| 14.3.6 | Summary of vital signs (Safety set) |
| 14.3.7 | Summary of change from baseline for vital signs (Safety set) |
| 14.3.8 | Summary of quantitative safety laboratory variables (Safety set) |
| 14.3.9 | Summary of qualitative safety laboratory variables (Safety set) |
| 14.3.10 | Summary of concomitant medication (Safety set) |

## 13 List of Listings

| 16.2.1 | Subject disposition |
|----------|---------------------------------------------|
| 16.2.1.1 | Screen failure subjects |
| 16.2.1.2 | Study completion status |
| 16.2.1.3 | Subject distribution in analysis population |
| 16.2.1.4 | Inclusion - Exclusion criteria |

# Lambda Therapeutic Research Ltd. Statistical Analysis Plan (SAP)

# Albendazole Tablets IP 400 mg

Version 00

| 16.2.1.5 | Inclusion criteria description |
|---|---|
| 16.2.1.6 | Exclusion criteria description |
| 16.2.2 | Protocol deviations |
| 16.2.3 | Subjects excluded from the analysis |
| 16.2.3.1 | Subjects excluded from the analysis (PK set) |
| 16.2.4 | Demographic data |
| 16.2.4.1 | Demographic data and baseline characteristics |
| 16.2.4.2 | Personal history |
| 16.2.4.3 | Medical and surgical history details |
| 16.2.4.4 | Physical examination |
| 16.2.4.5 | Medication history |
| 16.2.5 | Compliance and/or drug concentration data |
| 16.2.5.1 | Study drug administration |
| 16.2.5.2 | Compliance assessment |
| 16.2.5.3 | PK Sample collection |
| 16.2.5.4 | Concentration-time data for albendazole |
| 16.2.5.5 | Pharmacokinetic data for albendazole |
| 16.2.5.6 | Concentration-time data for albendazole sulfoxide |
| 16.2.5.7 | Pharmacokinetic data for albendazole sulfoxide |
| 16.2.7 | Adverse events (each subject) |
| 16.2.7.1 | Adverse events by severity, relationship to the study drug and by MedDRA term |
| 16.2.7.2 | Serious adverse events (if applicable) |
| 16.2.8 | Listing of individual laboratory measurements (by Subject) |
| 16.2.8.1 | Central laboratory tests |
| 16.2.8.2 | Safety laboratory analysis |
| 16.2.9 | Individual subject data listings |
| 16.2.9.1 | 12 Lead electrocardiogram |
| 16.2.9.2 | Chest x-ray |
| 16.2.9.3 | Body measurements |
| 16.2.9.4 | Vital signs |
| 16.2.9.5 | Urine drug scan and breath alcohol test |
| 16.2.9.6 | Lifestyle compliance assessment |
| 16.2.9.7 | Subjects date of visit |
| 16.2.9.8 | Unscheduled visit (if applicable) |
| 16.2.10 | Prior - concomitant medication |
| 14 List of Figures | |
| 14.2.4 | Figures of pharmacokinetic data |



| 14.2.4.1 | Mean plasma concentration vs. time curve for albendazole (Linear and Semi- |
|---|---|
| | log Plot) |
| 14.2.4.2 | Combined mean plasma concentration vs. time curve for albendazole (Linear and Semi-log Plot) |
| 14.2.4.3 | Mean (± SD) plasma concentration vs. time curve for albendazole (Linear and Semi-log Plot) |
| 14.2.4.4 | Median plasma concentration vs. time curve for albendazole (Linear and Semi-log Plot) |
| 14.2.4.5 | Median (range) plasma concentration vs. time curve for albendazole (Linear and Semi-log Plot) |
| 14.2.4.6 | Summary plot of individual plasma concentration vs time for albendazole (Linear and Semi-log Plot) |
| 14.2.4.7 | Mean plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |
| 14.2.4.8 | Combined mean plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |
| 14.2.4.9 | Mean (± SD) plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |
| 14.2.4.10 | Median plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |
| 14.2.4.11 | Median (range) plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |
| 14.2.4.12 | Summary plot of individual plasma concentration vs time for albendazole sulfoxide (Linear and Semi-log Plot) |
| 16.2.6 | Individual pharmacokinetic response data |
| 16.2.6.1 | Individual plasma concentration vs. time curve for albendazole (Linear and Semilog Plot) |
| 16.2.6.2 | Individual plasma concentration vs. time curve for albendazole sulfoxide (Linear and Semi-log Plot) |

#### 15 List of In-text Tables

- 1 Summary of Adverse Events
- 2 Summary of Adverse Events with System Organ Class

# 16 Statistical Outputs

| 16.1.9 | Documentation of statistical methods |
|---|---|
| 16.1.9.1 | Raw SAS output of intra-subject variability and SWR of Reference formulation for albendazole |
| 16.1.9.2 | Raw SAS output of ANOVA and BE for albendazole |
| 16.1.9.3 | Raw SAS output of intra-subject variability and SWR of Reference formulation for albendazole sulfoxide |
| 16.1.9.4 | Raw SAS output of ANOVA and BE for albendazole sulfoxide |
| 16.1.9.5 | Statistical Analysis Plan |

Note: Numbering in outputs may change depending on the inclusion/exclusion of the subjects considered for statistical analysis.



#### 17 References

- 1. ICH Harmonized Tripartite Guideline Statistical Principles for Clinical Trials (E9). Step 5 September 1998.
- 2. ICH Harmonized Tripartite Guideline Structure and Content of Clinical Study Reports (E3). Step 5 July 1996.
- 3. WHO Expert Committee on Specifications for Pharmaceutical Preparations. Fifty-fifth report (TR1033), annex 6: Multisource (generic) pharmaceutical products: guidelines on registeration requirements to establish interchangeability. World Health Organisation. 25 March 2021



### 18 Tables and Listings shells

14.1 Demographic Data

14.1.1 Demographic data and baseline characteristics (Randomized set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.1.1

Demographic data and baseline characteristics (Randomized set)

| | Statistics | TRTR<br>(N=xx) | RTRT<br>(N=xx) | Total<br>(N=xx) | p-value |
|---|---|---|---|---|---|
| Age (years) | n | XX | XX | XX | X.XXXX |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX.X | XX.X | XX.X | |
| | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X | |
| Gender | | | | | - |
| Male | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Female | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Race | | | | | |
| Asian | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | - |
| American Indian or Alaska Native | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Other | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Ethnicity | | | | | |
| Not Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | _ |
| Hispanic or Latino | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Not Reported | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Unknown | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x) | |
| Height (cm) | n | xx | xx | XX | x.xxxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX.X | XX.X | XX.X | |
| | Min, Max | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x | |

Project No. 0110-23 Version 00

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.1.1

Demographic data and baseline characteristics (Randomized set)

| | Statistics | TRTR<br>(N=xx) | RTRT<br>(N=xx) | Total<br>(N=xx) | p-value |
|---|---|---|---|---|---|
| Weight (kg) | n | XX | XX | XX | x.xxxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX.X | XX.X | XX.X | |
| | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x | |
| BMI (kg/m²) | n | xx | xx | xx | x.xxx |
| | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) | |
| | Median | XX.X | XX.X | XX.X | |
| | Min, Max | XX.X, XX.X | xx.x, xx.x | XX.X, XX.X | |

N = Number of subjects in safety set, n = Number of subjects in respective categories Note: Percentages are calculated based on the total number of subjects in each category. Treatment specification -> T = Test Product and R = Reference Product. p-value is calculated using an independent t-test. Reference Listings: 16.2.1.3, 16.2.4.1, 16.2.9.3

Output Generated on: DDMMMYYYY hh:mm

<Note: Repeat the same table as 14.1.2 for Safety set and 14.1.3 for PK set >

Project No. 0110-23 Version 00

14.1.4 Visit wise distribution of subjects (Randomized set)

Lambda Therapeutic Research Ltd. Confidential Project No. 0110-23

Table 14.1.4

Visit wise distribution of subjects (Randomized set)

| Visits | TRTR (N=xx) | RTRT<br>(N=xx) | Total (N=xx) |
|------------------|-------------|----------------|--------------|
| | n (%) | n (%) | n (%) |
| PERIOD 1 (Day-1) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PERIOD 2 (Day-1) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PERIOD 3 (Day-1) | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PERIOD 4 (Day-1) | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in safety set, n = Number of subjects in respective categories Note: Percentages are calculated based on the total number of subjects in each category. Treatment specification -> T = Test Product and R = Reference Product. Reference Listing: 16.2.1.3, 16.2.9.7

Output Generated on: DDMMMYYYY hh:mm

<Note: Repeat the same table as 14.1.5 for Safety set and 14.1.6 for PK set.>

Project No. 0110-23 Version 00

14.1.7 Summary of protocol deviations

Lambda Therapeutic Research Ltd.

Table No. 14.1.7
Summary of protocol deviations

Project No. 0110-23

| Protocol deviation | Type of Proto | Total | |
|-----------------------------------|---------------|-------|-------|
| FIOLOCOI deviación | Major | Minor | iotai |
| Subjects with protocol deviations | XX | XX | xx |
| At least one protocol deviation | xx | xx | xx |
| Dosing Related | xx | XX | XX |
| IMP Related | xx | xx | xx |
| Lab Related | xx | XX | XX |
| Others | xx | xx | xx |
| • | | | |

Reference Listing: 16.2.2

Output Generated on: DDMMMYYYY hh:mm

# **Project No. 0110-23** Version 00



#### 14.2 Pharmacokinetic Data 14.2.1 Plasma Albendazole Data

14.2.1.1 Summary statistics of pharmacokinetic parameters for albendazole

Lambda Therapeutic Research Ltd. Confidential Project No. 0110-23 The SAS System Version 9.4 Table No. 14.2.1.1 Sponsor: GSK Research & Development

Summary statistics of pharmacokinetic parameters for albendazole  $% \left( \frac{1}{2}\right) =\frac{1}{2}\left( \frac{1}{2}\right) +\frac{1}{2}\left( \frac{1}{2}\right) +\frac{1}{2}\left($ 

Albendazole Tablets IP 400 mg

| Measures | Tmax | Cmax | AUC0-t |
|---|---|---|---|
| | (unit) | (unit) | (unit) |
| Test Treatment-T | | | |
| N | XX | xx | XX |
| Mean | XX.XX | XX.XXX | xx.xxx |
| SD | XX.XXX | XX.XXXX | XX.XXXX |
| CV (%) | XX.X | XX.X | XX.X |
| Geometric Mean | XX.XX | XX.XXX | XX.XXX |
| Reference Treatment-R | | | |
| N | XX | XX | XX |
| Mean | XX.XX | XX.XXX | XX.XXX |
| SD | xx.xxx | XX.XXXX | xx.xxxx |
| CV (%) | xx.x | XX.X | XX.X |
| Geometric Mean | XX.XX | XX.XXX | XX.XXX |
| ANOVA p-value | | | |
| <br>ln-transformed Sequence | _ | x.xxxx | x.xxxx |
| Period | _ | X.XXXX | x.xxxx |
| Formulation | _ | X.XXXX | x.xxxx |
| D = + 1 = 1 = + (Q = = ) | | | |
| Participant (Sequence) Geometric Least Squares Means | _ | x.xxx | x.xxx |
| Geometric Least Squares Means | - | x.xxxx<br>xxxx.xxx | x.xxxx<br>xxxx.xxx |
| Geometric Least Squares Means | -<br>-<br>- | | |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea | -<br>-<br>ns(%)(T/R) | xxxx.xxx | xxxx.xxx |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea | -<br>-<br>ns(%)(T/R) | xxxx.xxx | xxxx.xxx |
| Geometric Least Squares Means ln-transformed Test-T | | xxxx.xxx<br>xxxx.xxx | xxxx.xxx<br>xxxx.xxx |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Means In-transformed Intra subject Variability of Referen | | xxxx.xxx<br>xxxx.xxx | xxxx.xxx<br>xxxx.xxx |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Means In-transformed Intra subject Variability of Referen In-transformed | <br>-<br>ce Formulati<br>- | xxxx.xxx<br>xxxx.xxx<br>xxx.x<br>on-R(%) | xxxx.xxx<br>xxxx.xxx<br>xxx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Means In-transformed Intra subject Variability of Referen | <br>-<br>ce Formulati<br>- | xxxx.xxx<br>xxxx.xxx<br>xxx.x<br>on-R(%) | xxxx.xxx<br>xxxx.xxx<br>xxx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea In-transformed Intra subject Variability of Referen In-transformed Within subject standard deviation of In-transformed | <br>-<br>ce Formulati<br>- | xxxx.xxx xxxx.xx xxx.x on-R(%) xx.x ormulation-R (SW | xxxx.xxx<br>xxxx.xx<br>xxx.x<br>xx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea In-transformed Intra subject Variability of Referen In-transformed Within subject standard deviation of In-transformed | <br>-<br>ce Formulati<br>- | xxxx.xxx xxxx.xx xxx.x on-R(%) xx.x ormulation-R (SW | xxxx.xxx<br>xxxx.xx<br>xxx.x<br>xx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea In-transformed Intra subject Variability of Referen In-transformed Within subject standard deviation of In-transformed 90% Confidence Interval (T Vs. R) In-transformed Lower | <br>-<br>ce Formulati<br>- | xxxx.xxx xxxx.xx xxx.x on-R(%) xx.x ormulation-R (SW | xxxx.xxx xxx.x xxx.x xx.x xx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea In-transformed Intra subject Variability of Referen In-transformed Within subject standard deviation of In-transformed 90% Confidence Interval (T Vs. R) In-transformed Lower Upper | <br>-<br>ce Formulati<br>- | xxxx.xxx xxxx.xxx xxx.x on-R(%) xx.x ormulation-R (SW xx.x | xxxx.xxx xxx.x xxx.x xxx.x xx.x xx.x |
| Geometric Least Squares Means In-transformed Test-T Reference-R Ratio of Geometric Least Squares Mea In-transformed Intra subject Variability of Referen In-transformed Within subject standard deviation of In-transformed 90% Confidence Interval (T Vs. R) In-transformed Lower | <br>-<br>ce Formulati<br>- | xxxx.xxx xxxx.xxx xxx.x on-R(%) xx.x ormulation-R (SW xx.x xx.x | xxxx.xxx xxx.xx xxx.x xx.x xx.x xx.x xx.x |

Output Generated on: DDMMMYYYY hh:mm

<Note: Repeat the same table as 14.2.2.1 for albendazole sulfoxide >



14.2.1.2 Pharmacokinetic parameters (untransformed) of albendazole for Test Product-T and Reference Product-R

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.2

| Pharmacokinetic parameters (untransformed) of albendazole for Test Product-T and Reference Product-R | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Tmax | (unit) | Cmax (unit) | | | A | UC0-t (uni | t) | AUC0-inf (unit) | | |
| Participants S | Sequence | Formu | ılation | Formulation | | | H | Formulation | 1 | Formulation | | |
| | | T | R | T | R | (T/R)% | T | R | (T/R)% | T | R | (T/R)% |
| 1001 | | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X |
| 1002 | | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X |
| | | | | • | • | • | • | | • | • | • | • |
| | | | | • | • | • | • | | • | • | • | • |
| | | • | • | | | | | | | | | |
| n | | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X | XX.XXX | XX.XXX | XX.X |
| N | | XX | XX | XX | XX | - | XX | XX | - | XX | XX | - |
| Mean | | XX.XX | XX.XX | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - |
| 95% CI of arit | hmetic | X.XX- | x.xx- | x.xxx- | x.xxx- | - | x.xxx- | x.xxx- | - | x.xxx- | x.xxx- | - |
| mean | | X.XX | X.XX | X.XXX | X.XXX | | X.XXX | X.XXX | | X.XXX | X.XXX | |
| SD | | XX.XXX | XX.XXX | XX.XXXX | XX.XXXX | - | XX.XXXX | XX.XXXX | - | XX.XXXX | XX.XXXX | - |
| Min | | XX.XX | XX.XX | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - |
| Median | 1 | XX.XX | XX.XXX | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - |
| Max | | XX.XX | XX.XX | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - |
| CV% | | XX.X | XX.X | XX.X | XX.X | - | XX.X | XX.X | - | XX.X | XX.X | - |
| Geometric Mean | | XX.XX | XX.XX | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - | XX.XXX | XX.XXX | - |
| 95% CI of geome | etric mean | X.XX-<br>X.XX | X.XX- | X.XXX- | X.XXX- | - | X.XXX- | X.XXX- | - | X.XXX- | X.XXX- | - |
| al a D | | | X.XX | X.XXX | X.XXX | | X.XXX | X.XXX | | X.XXX | X.XXX | |

Note: Repeat the same table as 14.2.2.2 for albendazole sulfoxide.>



14.2.1.2 Contd 1. Pharmacokinetic parameters (untransformed) of albendazole for Test Product-T and Reference Product-R

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.2 Contd.

Pharmacokinetic parameters (untransformed) of albendazole for Test Product-T and Reference Product-R

| | | AUC_%Extr | ap_obs (%) | Lambda | a_z (unit) | t1/2 (unit) | |
|---|---|---|---|---|---|---|---|
| Participants | Sequence | Formul | ation | Form | ulation | Formulation | |
| | | Т | R | T | R | T | R |
| 1001 | 1001 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| 1002 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| | | | | | • | | |
| | | | • | • | | • | |
| | | | • | • | | • | |
| n | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | N | | XX | XX | XX | XX | XX |
| N | Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% | 95% CI of | | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- |
| arithme | etic mean | X.XXX | x.xxx | X.XXX | X.XXX | X.XXX | x.xxx |
| | SD | | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX |
| ] | Min | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Med | Median | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| I | Max | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| | CV% | | XX.X | XX.X | XX.X | XX.X | XX.X |
| Geom | Geometric Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx |
| 95% CI of ge | 95% CI of geometric mean | | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- |
| | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |

<Note: Repeat the same table as 14.2.2.2 for albendazole sulfoxide.>



14.2.1.3 Individual Pharmacokinetic parameter (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

Lambda Therapeutic Research Ltd.

Confidential Table No. 14.2.1.3

Project No. 0110-23

Individual pharmacokinetic parameters (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

| | | | Tmax ( | (unit) | | | Cmax (ur | nit) | | AUC0-t (unit) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Participants | Participants Sequence | | Formu | lation | | | Formulat | ion | | Formulation | | | |
| | | T1 | T2 | R1 | R2 | T1 | T2 | R1 | R2 | T1 | T2 | R1 | R2 |
| 1001 | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 1002 | | xx.xx | XX.XX | XX.XX | XX.XX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | | | • | | | • | | • | | | • | | |
| | | • | • | • | • | • | • | • | • | • | • | • | |
| • | | | • | • | • | • | | | • | • | • | • | • |
| n | | XX.XX | XX.XX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| N | | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX | XX |
| Mea | an | XX.XX | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of a | arithmetic | x.xx- | x.xxx- | X.XX-X.XX | X.XX-X.XX | X.XXX- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- |
| mea | ın | X.XX | X.XXX | | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |
| SE | ) | xx.xxx | XX.XXXX | XX.XXX | XX.XXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX |
| Min | n | xx.xx | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Medi | ian | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Ma | X | xx.xx | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV | % | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Geometri | Geometric Mean | | XX.XXX | XX.XX | XX.XX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of § | 95% CI of geometric | | x.xxx- | X.XX-X.XX | X.XX-X.XX | X.XXX- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- |
| mea | n<br>1 | X.XX | X.XXX | 1 10 11 2 | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX |

<Note: Repeat the same table as 14.2.2.3 for albendazole sulfoxide >



14.2.1.3 Contd. Individual pharmacokinetic parameter (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.3 Contd.

Individual pharmacokinetic parameters (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

| | | | AUC0-inf | (unit) | | AUC_%Extrap_obs (%) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Participants | Sequence | | Formulatio | on | | Formulation | | | |
| | | T1 | T2 | R1 | R2 | T1 | T2 | R1 | R2 |
| 1001 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 1002 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | | | • | • | • | | • | • | |
| n | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | N | | XX | XX | XX | XX | XX | XX | XX |
| | Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CL c | 95% CI of arithmetic mean | | X.XXX- | X.XXX- | x.xxx- | x.xxx- | X.XXX- | x.xxx- | x.xxx-x.xxx |
| 7570 61 6 | | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | |
| | SD | | XX.XXXX | XX.XXXX | XX.XXXX | xx.xxxx | XX.XXXX | XX.XXXX | XX.XXXX |
| | Min | | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Median | | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Max | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Geomet | Geometric Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CL | 95% CI of geometric mean | | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | X.XXX-X.XXX |
| 9370 CT C | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | |

<Note: Repeat the same table as 14.2.2.3 for albendazole sulfoxide >

14.2.1.3 Contd. Individual pharmacokinetic parameter (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.3 Contd.

Individual pharmacokinetic parameters (untransformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

| | Sequence | | Lambda | a_z (unit) | | t1/2 (unit) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Participants | | | Form | ulation | | Formulation | | | |
| | | T1 | T2 | R1 | R2 | T1 | T2 | R1 | R2 |
| 1001 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 1002 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| | | • | • | • | | • | • | • | |
| n | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| N | N | | XX | XX | XX | XX | XX | XX | XX |
| Mear | Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of arithmetic mean | | X.XXX- | X.XXX- | X.XXX- | x.xxx- | x.xxx- | X.XXX- | x.xxx- | x.xxx-x.xxx |
| | 7570 CI of artifificate mean | | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | |
| SD | SD | | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX |
| Min | Min | | XX.XXX | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| Median | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Max | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Geometric | Geometric Mean | | XX.XXX | XX.XXX | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of geon | netric mean | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | x.xxx- | X.XXX-X.XXX |
| 7570 CI 01 gcon | ileti ie ilieali | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | X.XXX | |

<Note: Repeat the same table as 14.2.2.3 for albendazole sulfoxide >
14.2.1.4 Pharmacokinetic parameters (untransformed) of data excluded from statistical analysis for albendazole (if applicable)

Lambda Therapeutic Research Ltd.

Project No. 0110-23

Table No. 14.2.1.4


Pharmacokinetic parameters (untransformed) of data excluded from statistical analysis for albendazole

| Participants | Period | Sequence | Formulation | Tmax (unit) | Cmax<br>(unit) | AUC0-t<br>(unit) | AUC0-inf<br>(unit) | AUC_%Extrap_obs (%) | Lambda_z<br>(unit) | t1/2<br>(unit) |
|---|---|---|---|---|---|---|---|---|---|---|
| 1001 | | | | XX.XXX | XX.XXX | xx.xxx | XX.XXX | xx.xxx | xx.xxx | xx.xx |
| 1002 | | | | xx.xxx | xx.xxx | xx.xxx | XX.XXX | XX.XXX | xx.xxx | xx.xx |
| | | | | | | • | • | | • | |
| | | | | | | • | • | • | • | |
| | | | | | | | | • | | |
| n | | | | xx.xxx | xx.xxx | xx.xxx | XX.XXX | xx.xxx | xx.xxx | xx.xx |

<Note: Repeat the same table as 14.2.2.4 for albendazole sulfoxide.>



14.2.1.5 Pharmacokinetic parameters (In-transformed) of albendazole for Test Product-T and Reference Product-R

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.5

Pharmacokinetic parameters (In-transformed) of albendazole for Test Product-T and Reference Product-R

| | | Cma | ax | Α | AUC0-t |
|---|---|---|---|---|---|
| Participants | Sequence | Formul | ation | Formulation | |
| | | T | R | T | R |
| 1001 | | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 1002 | | XX.XXX | XX.XXX | xx.xxx | XX.XXX |
| n | | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| N | | XX | XX | XX | XX |
| Mean | | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of arithr | netic mean | X.XXX-X.XXX | x.xxx-x.xxx | x.xxx-x.xxx | X.XXX-X.XXX |
| SD | | XX.XXXX | XX.XXXX | XX.XXXX | XX.XXXX |
| Min | | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Media | n | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| Max | | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| CV% | | XX.X | XX.X | XX.X | XX.X |
| Geometric M | ean | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of geom | etric mean | X.XXX-X.XXX | X.XXX-X.XXX | X.XXX-X.XXX | X.XXX-X.XXX |

<Note: Repeat the same table as 14.2.2.5 for albendazole sulfoxide.>



14.2.1.6 Individual Pharmacokinetic parameter (In-transformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table No. 14.2.1.6

Individual pharmacokinetic parameters (In-transformed) of albendazole for Test Product-T1 (first administration), Test Product-T2 (second administration), Reference Product-R1 (first administration) and Reference Product-R2 (second administration)

| | | Cr | Cmax (unit) | | | AUC0-t (unit) | | | |
|---|---|---|---|---|---|---|---|---|---|
| Participants | Sequence | Fo | rmulation | | | Formulation | | | |
| | | T1 | T2 | R1 | R2 | T1 | T2 | R1 | R2 |
| 1001 | | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | xx.xxx | XX.XXX |
| 1002 | | XX.XXX | xx.xxx | xx.xxx | xx.xxx | xx.xxx | xx.xxx | XX.XXX | XX.XXX |
| | | | • | • | • | | • | | |
| • | | • | • | • | • | • | • | • | |
| | | | • | • | • | • | • | • | • |
| n | | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | N | XX | XX | XX | XX | XX | XX | XX | XX |
| ı | Mean | XX.XXX | xx.xxx | xx.xxx | xx.xxx | xx.xxx | xx.xxx | XX.XXX | XX.XXX |
| 95% CI of a | arithmetic mean | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx |
| | SD | xx.xxxx | xx.xxx | xx.xxx | xx.xxx | xx.xxx | xx.xxxx | xx.xxx | XX.XXXX |
| | Min | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| M | Iedian | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | Max | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| Geom | etric Mean | XX.XXX | XX.XXX | xx.xxx | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX |
| 95% CI of § | geometric mean | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | x.xxx-x.xxx | X.XXX-X.XXX | x.xxx-x.xxx | x.xxx-x.xxx |

<Note: Repeat the same table as 14.2.2.6 for albendazole sulfoxide.>

### 14.2.1.7 Plasma concentration of albendazole for Test Product-T1 (first administration)

Lambda Therapeutic Research Ltd.

### Confidential

Project No. 0110-23

| Tal | ble | 14.2. | 1.7 |
|-----|-----|-------|-----|

| | | oncentration of<br>oduct-T1 (first a | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Time | | Participan | ts | | N | Mean | SD | Min | Median | Max | CV% | Geometric |
| (unit) | | Concentration | (unit) | | | | | | | | | Mean |
| | 1001 | 1002 | | n | | | | | | | | |
| $T_1$ | xx.xxx | XX.XXX | | XX.XXX | XX | x.xxx | x.xxxx | x.xxx | x.xxx | X.XXX | X.X | x.xxx |
| $T_2$ | XX.XXX | XX.XXX | | XX.XXX | XX | x.xxx | x.xxxx | x.xxx | x.xxx | x.xxx | X.X | x.xxx |
| • | • | • | | • | | • | • | • | • | • | • | |
| • | • | • | • | • | • | • | • | • | ٠ | • | • | |
| | | | | • | | • | | | • | • | • | |
| | | | | | | | | | • | • | • | |
| | | | | • | | • | | | • | • | • | |
| $T_{i}$ | XX.XXX | XX.XXX | • | XX.XXX | XX | X.XXX | X.XXXX | X.XXX | X.XXX | X.XXX | X.X | X.XXX |

*Note: Here*  $T_i$  ( $i = 1, 2, \ldots, n$ ) denotes the time points at which blood sample has been taken

<sup>&</sup>lt;Note 1: Repeat the same table as 14.2.1.8 for Test Product-T2 (second administration), 14.2.1.9 for Reference Product-R1 (first administration) and 14.2.1.10 for Reference Product-R2 (second administration) of albendazole.>

<sup>&</sup>lt;Note 2: Repeat the same table as 14.2.2.7 for Test Product-T1 (first administration), 14.2.2.8 for Test Product-T2 (second administration), 14.2.2.9 for Reference Product-R1 (first administration) and 14.2.2.10 for Reference Product-R2 (second administration) of albendazole sulfoxide.>

14.2.1.11 Plasma concentration of data excluded from statistical analysis for albendazole (if applicable)

Lambda Therapeutic Research Ltd.

Table 14 2 1 11

Project No. 0110-23

| | | 1able 14.2.1.11 | | |
|---|---|---|---|---|
| | Plasma concentration of | Plasma concentration of data excluded from statistical analysis for albendazole | | |
| | | Participants | | |
| Time (h) | | Concentration | (unit) | |
| Time (h) | 1001 | 1002 | | n |
| | Period | Period | | Period |
| | Formulation | Formulation | | Formulation |
| $T_1$ | XX.XXX | XX.XXX | | XX.XXX |
| $T_2$ | XX.XXX | XX.XXX | | XX.XXX |
| | | • | • | |
| | | • | • | |
| • | | • | • | |
| • | | • | • | |
| <u>·</u> | | | • | |
| $T_{i}$ | XX.XXX | XX.XXX | | XX.XXX |

*Note: Here*  $T_i$  ( $i = 1, 2, \ldots, n$ ) denotes the time points at which blood sample has been taken.

<sup>&</sup>lt;Note: Repeat the same table as 14.2.2.12 for albendazole sulfoxide.>

## 14.2.3 Actual time points used for pharmacokinetic evaluation

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.2.3

Actual time points used for pharmacokinetic evaluation

| Participants | Period | Time Point<br>(unit) | Difference in<br>Minutes | Difference in Hour | Actual Time of Collection (unit) |
|---|---|---|---|---|---|
| 1001 | | x.xxx | | x.xxx | x.xxx |
| 1002 | | x.xxx | | x.xxx | x.xxx |
| • | | • | | | |
| | | • | | • | |
| • | | • | | • | |
| • | | • | | • | |
| • | | • | | • | |
| • | | • | | • | |
| • | | • | | • | |
| • | | • | | • | • |
| n | | x.xxx | | X.XXX | x.xxx |

## 14.3 Safety Data

14.3.1 Overall summary of treatment emergent adverse events (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.1

| | Test Treatment-T | Reference Treatment-R | Total | |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | p-valu |
| | n (%) e | n (%) e | n (%) e | |
| At least one TEAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | x.xxx |
| At least one TEAE leading to discontinuation | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | X.XXX |
| At least one TESAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | _ |
| Assessment of intensity | | | | _ |
| Mild | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Moderate | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Severe | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Seriousness criteria | | | | - |
| Congenital Anomaly/Birth Defect | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Hospitalization or prolongation of existing | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| hospitalization | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Result in persistent or Significant | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Disability/incapacity | AA (AA.A) AA | AA (AA.A) AA | AA (AA.A) AA | |
| Life threatening | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Abnormal pregnancy outcomes | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Death | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Other Medically Important Event | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Relationship to Study Treatment | | | | _ |
| Related | | | | |
| Certain | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Probable/Likely | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Possible | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Not Related | | | | |
| Unlikely | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Conditional/Unclassified | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |



Lambda Therapeutic Research Ltd.

Confidential Table 14.3.1

Project No. 0110-23

Overall summary of treatment emergent adverse events (Safety set)

| | Test Treatment-T | Reference Treatment-R | Total | |
|---|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) | p-value |
| | n (%) e | n (%) e | n (%) e | |
| Unassessable/Unclassifiable | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Unrelated | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Action Taken with Study Treatment | | | | _ |
| Dose Increased | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Dose Not Changed | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Dose Reduced | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Drug Interrupted | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Drug Withdrawn | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Not Applicable | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Unknown | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Outcome | | | | _ |
| Not Recovered/Not Resolved | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Recovering/resolving | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Recovered/Resolved | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Recovered/Resolved With Sequelae | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Stable | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Change in severity | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Fatal | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Converted to SAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Unknown | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |
| Death | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | |

N = Number of subjects in respective treatment population.

Reference Listing: 16.2.7.1

n = Number of subjects in respective categories; e = Number of events.

Percentages are based on the number of subjects allocated to each category.

P-value is calculated based on a chi-square test. If any cell has expected counts less than 5, then the Fisher's exact test is used instead.



14.3.2 Summary of treatment emergent adverse events by system organ class and preferred term (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.2

Summary of treatment emergent adverse events by system organ class and preferred term (Safety set)

| | Test Treatment-T | Reference Treatment-R | Total |
|---|---|---|---|
| System Organ Class | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | n (%) e | n (%) e | n (%) e |
| Subjects with At least one TEAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • | | | |
| • | | | |
| System Organ Class 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Etc. | | | |

N = Number of subjects in respective treatment population.

n = Number of subjects in respective categories; e = Number of events.

Percentages are based on the number of subjects allocated to each category.

Each subjects is counted at the most once within each PT.

Adverse Events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version xx

Reference Listing: 16.2.7.1

Project No. 0110-23 Version 00

14.3.3 Summary of treatment emergent adverse events by relationship to study drug and system organ class and preferred term (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.3

Summary of treatment emergent adverse events by relationship to study drug and system organ class and preferred term (Safety set)

| System Organ Class<br>Preferred Term | (N= | atment-T<br>xxx)<br>%) e | (N= | Treatment-R<br>=xx)<br>%) e | Total<br>(N=xx)<br>n (%) e | |
|---|---|---|---|---|---|---|
| | Related | Not-Related | Related | Not-Related | Related | Not-Related |
| Subjects with At least one TEAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| System Organ Class 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| ·<br>· | | | | | | |
| | xx (xx.x) xx | xx (xx.x) xx | () | () | () | xx (xx.x) xx |
| System Organ Class 2 | , , | , | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | • |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Etc. | | | | | | |

N = Number of subjects in respective treatment population.

n = Number of subjects in respective categories; e = Number of events.

Percentages are based on the number of subjects allocated to each category.

Each subject is counted at most once within each PT.

Adverse Events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version xx

Reference Listing: 16.2.7.1



14.3.4 Summary of treatment emergent adverse events by severity grade and system organ class and preferred term (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.4

Summary of treatment emergent adverse events by severity grade and system organ class and preferred term (Safety set)

| | Test Treatment-T | Reference Treatment-R | Total |
|---|---|---|---|
| System Organ Class | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | n (%) e | n (%) e | n (%) e |
| Subjects with At least one TEAE | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Mild | | | |
| System Organ Class 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| • | | | |
| • | | | |
| System Organ Class 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 1 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Preferred Term 2 | xx (xx.x) xx | xx (xx.x) xx | xx (xx.x) xx |
| Etc. | | | |

N = Number of subjects in respective treatment population.

n = Number of subjects in respective categories; e = Number of events.

Percentages are based on the number of subjects allocated to each category.

Each subject is counted at most once within each PT.

Adverse Events are coded using Medical Dictionary for Regulatory Activities (MedDRA) version xx Reference Listing: 16.2.7.1

Project No. 0110-23



# Lambda Therapeutic Research Ltd. Statistical Analysis Plan (SAP) Albendazole Tablets IP 400 mg

14.3.5 Summary of subject disposition

Lambda Therapeutic Research Ltd.


Table 14.3.5

Summary of subject disposition

| | TRTR | RTRT | Total |
|---------------------------------|-----------|-----------|-----------|
| | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (응) | n (%) |
| Subjects Randomized | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects included in Safety set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects included in PK set | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects who completed study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subjects who discontinued study | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason for discontinuing study | | | |
| Reason 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Reason 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in safety set, n = Number of subjects in respective categories Note: Percentages are calculated based on the total number of subjects in each category. Treatment specification  $\rightarrow$  T = Test Product and R = Reference Product. Reference Listing: 16.2.1.2

Output Generated on: DDMMMYYYY hh:mm

<Note for programmers: Reason for discontinued should be in descending order i.e., highest reported reasons should come first.>



14.3.6 Summary of vital signs (Safety set)

Lambda Therapeutic Research Ltd.

#### Confidential

Project No. 0110-23

Table 14.3.6

Summary of vital signs (Safety set)

| Parameters<br>(Unit) | Visit (Day) | Time Point | Statistics | TRTR (N=xx) | RTRT<br>(N=xx) | Total<br>(N=xx) | p-value |
|---|---|---|---|---|---|---|---|
| Pulse rate (beats/min) | Screening | | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | x.xxx |
| | Assessment<br>Visit X | Time Point 1 | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | x.xxxx |
| | | Time Point 2 | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | x.xxxx |
| | Assessment<br>Visit Y | Time Point 1 | n<br>Mean (SD)<br>Median<br>Min, Max | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | xx<br>xx.x (xx.xx)<br>xx.x<br>xx.x, xx.x | x.xxxx |
| Etc. | Etc. | Etc. | , | . , | . , | . , | |

N = Number of subjects in safety set, n = Number of subjects in respective categories

P-value is calculated using an independent t-test.

Treatment specification  $\rightarrow$  T = Test Product and R = Reference Product.

Reference Listing: 16.2.9.4

Output Generated on: DDMMMYYYY hh:mm

<Note for programmers: This table will continue for vital parameters like Systolic Blood Pressure (mmHg), Diastolic Blood Pressure (mmHg), Oral Body Temperature (°F), etc.>



14.3.7 Summary of change from baseline for vital signs (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.7

| Parameters | TT: '. (D.) | m: | | TRTR | RTRT | Total |
|---|---|---|---|---|---|---|
| (Unit) | Visit (Day) | Time Point | Statistics | (N=xx) | (N=xx) | (N=xx) |
| Diastolic Blood<br>Pressure (mmHg) | Assessment<br>Visit X | Time Point 1 | n | xx | xx | xx |
| | | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | | Median | xx.x | XX.X | XX.X |
| | | | Min, Max | XX.X, XX.X | XX.X, XX.X | XX.X, XX.X |
| | | Time Point 2 | n | XX | XX | xx |
| | | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Min, Max | xx.x, xx.x | XX.X, XX.X | xx.x, xx.x |
| | Assessment<br>Visit Y | Time Point 1 | n | xx | xx | xx |
| | | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | | Median | XX.X | XX.X | XX.X |
| | | | Min, Max | xx.x, xx.x | xx.x, xx.x | XX.X, XX.X |
| Etc. | Etc. | Etc. | | | | |

N = Number of subjects in safety set, n = Number of subjects in respective categories Change from Baseline (CFB) = Post Baseline assessment - Baseline assessment (0.00 Hrs Pre-Dose). Treatment specification -> T = Test Product and R = Reference Product. Reference Listing: 16.2.9.4

Project No. 0110-23



# Lambda Therapeutic Research Ltd. Statistical Analysis Plan (SAP) Albendazole Tablets IP 400 mg

14.3.8 Summary of quantitative safety laboratory variables (Safety set)

Lambda Therapeutic Research Ltd.


Table 14.3.8

Summary of quantitative safety laboratory variables (Safety set)

| Parameters | Visit | Statistics | TRTR | RTRT | Total |
|---|---|---|---|---|---|
| (Unit) | VISIC | Statistics | (N=xx) | (N=xx) | (N=xx) |
| Hemoglobin<br>(g/dL) | Screening | n | XX | XX | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | xx.x |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Assessment Visit X | n | xx | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | xx.x | xx.x | XX.X |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| | Assessment Visit Y | n | xx | xx | xx |
| | | Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| | | Median | XX.X | XX.X | XX.X |
| | | Min, Max | xx.x, xx.x | xx.x, xx.x | xx.x, xx.x |
| Etc. | Etc. | | | | |

N = Number of subjects in safety set, n = Number of subjects in respective categories

Treatment specification  $\rightarrow$  T = Test Product and R = Reference Product.

Quantitative data values observed out of limit of quantification are adjusted to quantification limits for descriptive statistics. In case of repeat sample collection latest result has been considered for the analysis.

Reference Listings: 16.2.8.1

Output Generated on: DDMMMYYYY hh:mm

<Note to Programmer: This table will continue for all other Laboratory parameters and some additional test.>

Project No. 0110-23



# Lambda Therapeutic Research Ltd. **Statistical Analysis Plan (SAP)** Albendazole Tablets IP 400 mg

14.3.9 Summary of qualitative safety laboratory variables (Safety set)

Lambda Therapeutic Research Ltd.


Table 14.3.9

Summary of qualitative safety laboratory variables (Safety set)

| Parameters (Unit) | Visit | Result | Statistics | TRTR<br>(N=xx) | RTRT<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|---|---|---|
| HBsAg | Screening | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Assessment Visit X | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | Assessment Visit Y | xxx | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| | | XXX | n (%) | xx (xx.x) | xx (xx.x) | xx (xx.x |
| Etc. | Etc. | | | | | |

N = Number of subjects in safety set, n = Number of subjects in respective categories Note: Percentages are calculated based on the total number of subjects in each category.

Treatment specification  $\rightarrow$  T = Test Product and R = Reference Product.

In case of repeat sample collection latest result has been considered for the analysis.

Reference Listing: 16.2.8.1

Output Generated on: DDMMMYYYY hh:mm

<Note to Programmer: This table will continue for all other Laboratory parameters and some additional test.>



14.3.10 Summary of concomitant medication (Safety set)

Lambda Therapeutic Research Ltd.


Project No. 0110-23

Table 14.3.10

Summary of concomitant medication (Safety set)

| | TRTR | RTRT | Total |
|---|---|---|---|
| | (N=xx)<br>n (%) | (N=xx)<br>n (%) | (N=xx)<br>n (%) |
| At least one concomitant medication | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Medication 3 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Etc. | xx (xx.x) | xx (xx.x) | xx (xx.x) |

N = Number of subjects in safety set, n = Number of subjects in respective categories Note: Percentages are calculated based on the total number of subjects in each category. Treatment specification  $\rightarrow$  T = Test Product and R = Reference Product. Reference Listing: 16.2.10

## **In-text tables**

Table 1: Summary of Adverse events

| Adverse events (as per MedDRA<br>PT - Version xxx) | Albendazole tablets IP<br>400 mg<br>Test (T) | Albendazole 400 mg<br>tablets<br>Reference (R) | Total |
|---|---|---|---|
| XXXXXXXX | X | X | х |
| XXXXXXXX | X | X | X |
| otal | X | X | X |

Table 2: Summary of Adverse Events with System Organ Class

| System Organ Class | MedDRA (PT)<br>(Version xxx) | Albendazole tablets IP<br>400 mg<br>Test (T) | Albendazole 400 mg<br>tablets<br>Reference (R) | No. of events |
|---|---|---|---|---|
| XXXXXXXXX | XXXXXXXX | X | X | X |
| XXXXXXXX | XXXXXXXX | X | X | X |
| XXXXXXXX | XXXXXXXX | X | X | X |
| XXXXXXXX | XXXXXXXX | X | X | x |
| XXXXXXXX | XXXXXXXX | X | X | X |
| XXXXXXXX | XXXXXXXX | X | X | x |
| XXXXXXXXX | XXXXXXXX | X | X | x |
| XXXXXXXX | XXXXXXXX | X | X | x |
| XXXXXXXX | XXXXXXXX | X | X | X |
| XXXXXXXX | XXXXXXXX | X | X | x |
| XXXXXXXX | XXXXXXXX | X | X | x |
| Total | | X | X | X |



## Listings

16.2.1 Subject disposition

| 16.2.1.1 Sc | reen fail | ure subje | cts | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Screening<br>No. | Date o | | Subject Study<br>upletion Statu | | for Screen | ', 'Physician on<br>ndrawal by subj<br>please specif | ect', | - | |
| Screenin<br>No. | _ | ate of<br>reening | inclusion | , | ment of<br>criteria or<br>please specif | 'Death', Date<br>Death | of | _ | |
| 16.2.1.2 St | tudy compl | letion sta | atus | | | | | | |
| Subject<br>no. | Sequence | _ | ct Study<br>ion Status | | Completion o | te of last dose<br>drug administr | | Reason<br>Discontin | |
| Subject<br>no. | Sequence | | er', 'Physicia<br>Subject', <b>'</b> Adv | | | n-fulfilment of<br>eria or Protoco | | , | If 'Death',<br>Date of Death |
| 16.2.1.3 St | ubject dis | stribution | n in analysis | population | | | | | |
| Subject r | no. Sequ | uence | Subjects inc<br>Randomize | | Subjects i<br>Safet | Subjects in in PK s | | | |
| 16.2.1.4 In | nclusion - | - Exclusio | on criteria | | | | | | |
| Subject no. | Sequence | | e subject mee<br>usion criteri | | o, Mark the I<br>ion number(s | Does the su<br>any exclusio | _ | • | Mark the EXCLUSIC |



| 16.2.1.5 I | inclusion c | riteria d | lescription | | | | | |
|---|---|---|---|---|---|---|---|---|
| Со | de | Ir | nclusion criteri | la descriptio | on | | | |
| 16.2.1.6 E | Exclusion c | riteria d | lescription | | | | | |
| Со | de | Εz | clusion criteri | la descriptio | on | | | |
| 16.2.2 Pro | tocol devia | ations | | | | | | |
| Subject<br>no. | Sequence | Visit<br>No. | Date of deviati<br>Occurrence | ion Protoc<br>Sectio | | | | |
| Subject no. | Sequence | Visit<br>No. | Type<br>(Major/Minor) | Reason for deviation | Description<br>of the<br>Deviation | Corrective<br>Action | Preventive<br>Action | Impact<br>Assessment |
| | • | • | available data from the analysis | the source.> | | | | |
| 16.2.3.1 S | Subjects exc | cluded fr | om the analysis | (PK set) | | | | |
| Subject | No. | Period | Reason | | | | | |
| | | | | <del></del> | | | | |



16.2.4 Demographic data

16.2.4.1 Demographic data and baseline characteristics

| Screening Subject no. no. Sequence Sequence Sequence Sequence (Screening) Date of Informed consent form consent form signed signed (Study Specific) | Date of Age<br>Birth (Years) | Gender | Ethnicity | Race | If Other,<br>please<br>specify |
|---|---|---|---|---|---|
|---|---|---|---|---|---|

< Note for programmers: This listing will be created on Randomized set.>

### 16.2.4.2 Personal history

| Subject | Sequence | Personal history assessment | Reproductive |
|---------|----------|-----------------------------|--------------|
| no. | sequence | done for female subject? | status |

### 16.2.4.3 Medical and surgical history details

| Subject<br>no. | Sequence | Visit | Nature of condition | Medical/Surgical<br>history term | Medical/Surgical<br>history code |
|---|---|---|---|---|---|

| Subject<br>no. | Sequence | Visit | Start<br>date | End<br>date | Ongoing |
|----------------|----------|-------|---------------|-------------|---------|

### 16.2.4.4 Physical examination

| Subject no. | Sequence | Visit | Date of assessment | Body<br>System | Result | Specify if<br>Abnormal<br>CS/Not Done | Any New clinically significant abnormality finding or worsening of condition since last assessment? |
|---|---|---|---|---|---|---|---|

| Subject<br>no. | Sequence | Visit | If yes, please<br>select body System | If yes, please specify abnormality |
|---|---|---|---|---|



| 16.2.4.5 | Medication | history |
|----------|------------|---------|
|----------|------------|---------|

| Subject no. | Sequence | Subject taken any medication from 14 days prior to dosing of period I? |
|---|---|---|

16.2.5 Compliance and drug concentration data

16.2.5.1 Study drug administration

| Subject no. | Sequence | Visit | Study drug<br>administration<br>performed? | Date of study drug administration | Time of Study<br>drug<br>administration | Mouth check<br>done after<br>dosing? | If 'No',<br>then<br>specify | Any deviation during dosing? | If 'Yes',<br>please<br>specify |
|---|---|---|---|---|---|---|---|---|---|
|---|---|---|---|---|---|---|---|---|---|

#### 16.2.5.2 Compliance assessment

| Subject | t Seguence Visit | Has the subject been compliant to | If 'No', then | Has the subject been compliant to all post dose compliance criteria? | If No, then | |
|---|---|---|---|---|---|---|
| no. | bequence | VISIC | all pre dose compliance criteria?: | specify | all post dose compliance criteria? | specify |

#### 16.2.5.3 PK sample collection

| Subject Sequence | Visit | Time | Actual Date of PK | Actual Time of PK | Any | If 'Yes', please |
|---|---|---|---|---|---|---|
| no. Sequence | VISIL | point | sample collection | sample collection | Deviation? | specify |

#### 16.2.5.4 Concentration-time data for albendazole

| Participant | Comiondo | Period | Formulation | Form | Schedule Time | Actual Time | Concentration |
|---|---|---|---|---|---|---|---|
| raiticipant | Sequence | reliou | | FOLIII | (h) | (h) | (unit) |

Programming note: Similar listing will be generated for albendazole sulfoxide as 16.2.5.6.

#### 16.2.5.5 Pharmacokinetic data for albendazole

| Participant Sequence | Period | Formulation | Form | Tmax | Cmax | AUC0-t | AUC0-inf | AUC_%Extrap_obs | Lambda_z | t1/2 |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | (h) | (unit) | (unit) | (unit) | _ (응) | (unit) | (unit) |

Programming note: Similar listing will be generated for albendazole sulfoxide as 16.2.5.7.



16.2.7 Adverse events (each subject)

16.2.7.1 Adverse events by severity, relationship to the study drug and by MedDRA term

| Subject no. | Treatment | Adverse<br>event term | Adverse<br>Event Cod | Start<br>e date | . Start<br>Time | | End<br>time | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject no. | Treatment | Assessment intensit | of<br>advers | this<br>e event<br>ous? | specify | ous, Please<br>seriousnes<br>iteria | s t | lationship<br>to Study<br>reatment | Take<br>S | ction<br>en with<br>tudy<br>atment | Outcor | me treatmer | omitant<br>nt/Therapy<br>ven |
| Subject no. | Treatment | Preferred<br>Term | Preferred<br>Term code | System<br>Organ<br>Class | Lowest<br>Level<br>Term | Lowest<br>Level<br>Term Code | Hic<br>Lev<br>Ter | el High | Level<br>Code | High I<br>Group | rever | High Level<br>Group Term<br>Code | - |
| | - 3 | having an acrese events | | | uded in t | this listin | ıg. | | | | | | - |
| Subject no. | Treatment | Adverse<br>event term | Adverse<br>Event Cod | Start<br>e date | Start<br>Time | | End<br>time | | | | | | |
| Subject no. | Treatment | Preferred<br>Term | Preferred<br>Term code | System<br>Organ<br>Class | Lowest<br>Level<br>Term | Lowest<br>Level<br>Term Code | Hic<br>Lev<br>Ter | el High | Level<br>Code | High I<br>Group | reдет | High Level<br>Group Term<br>Code | _ |

Note: Only subjects having serious adverse events are included in this listing.



16.2.8 Listing of individual laboratory measurements (by Subject)

< Note for programmers: This listing will be created on Randomized set.>

16.2.8.1 Central laboratory tests

| | Laboratory Test group | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Subject<br>no. | Sequence | Visit | Date of sample collection | Time of sample collection | Laboratory<br>Test | Unit | Laborator<br>range -<br>Minimum | y Laboratory<br>range -<br>Maximum | Laboratory<br>Results | Flagging<br>(L/H/A/N) |
| 16.2.8.2 | Safety Lab | oratory | analysis | | | | | | | |
| Subject no. | Sequence | Visit | Date of sa<br>collecti | | of sample<br>lection | Specimen<br>Type | - | | | |
| Subject no. | Sequence | Visit | Panel<br>Name | Overall<br>Interpretatio | If Abno | - 1 | eat sample<br>status | If 'Other', then specify | -<br>- | |
| | dividual s | 3 | data listings<br>ardiogram | ; | | | | | | |
| Subject no. | Sequence interpretation - | | | | | | | | | |
| 6.2.9.2 | Chest x-ra | У | | | | | | | | |
| Subject no. | Sequence | Visit | Date o | Int | cerpretation | | bnormal CS, ase specify | | | |
| 16.2.9.3 | Body measu | rements | | | | | | | | |
| Subject | no. Sequ | ience | Height(cm) | Weight (Kgs) | BMI(kg/m²) | <u> </u> | | | | |



Subject

no.

Sequence

# Lambda Therapeutic Research Ltd. Statistical Analysis Plan (SAP) Albendazole Tablets IP 400 mg

Reason for

unscheduled

visit

Date of

unscheduled

visit

16.2.9.4 Vital signs

| Subject<br>no. | Sequenc | e Visit | Time<br>Point | Date of measurement | Time of measurement | Systolic blood<br>pressure | Diastolic blood<br>pressure | |
|---|---|---|---|---|---|---|---|---|
| Subject no. | Sequenc | e Visit | Radia<br>pulse | - | ry Body<br>temperatu | re Interpretation | If Abnormal CS, please specify | CFB |
| Change fr | om Basel | ine (CFB) | = Post | Baseline asse | essment - Basel | ine assessment (0 | 0.00 Hrs Pre-Dose) | |
| 16.2.9.5 | Urine dr | ıg scan a | and breat | th alcohol tes | st | | | |
| Subject<br>no. | Sequenc | e Visit | Date<br>assess | | drug<br>esult alcoh | eath<br>ol test<br>sult | | |
| _ | | | assess | ment scan r | drug<br>esult alcoh | ol test | | |
| no. | Lifestyl | e complia | assess | ment scan r essment Subject foll | drug<br>esult alcoh | ol test sult nstruction of | If "No" then specify | |
| no. | Lifestyl<br>no. Sec | e complia | assess | ment scan r essment Subject foll | drug alcoh re | ol test sult nstruction of | If "No" then specify | |

If Other,

please

specify

Activity

Name

If any abnormal clinically

significant findings, then

provide details



16.2.10 Prior - Concomitant medication

| Subject no. | Sequence | Medication<br>Name or<br>Therapy | Medication<br>Code | Indication code | Indication | Dose per administration | Unit | If 'Other' (Unit), please specify | ·<br>- |
|---|---|---|---|---|---|---|---|---|---|
| Subject no. | Sequence | Frequency | If 'Ot<br>(Freque<br>please s | ncy), | Route ( | If 'Other'<br>Route), please<br>specify | Start<br>date | End date | Ongoing |